CLINICAL TRIAL: NCT00354354
Title: Bronchodilator Effect on O2 Deficit and V'O2 Kinetics During Moderate Intensity Exercise in Normoxemic COPD.
Brief Title: Bronchodilators and Oxygen Kinetics With Exercise in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Dr. Denis O'Donnell, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DMED-926-06
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Combivent; Exercise; Bronchodilator; Kinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Combivent
  Interventions: Drug: Combivent
- 2 (Placebo Comparator): Saline Solution (0.9% NaCl)
  Interventions: Drug: Combivent

INTERVENTIONS:
Drug: Combivent — Nebulized Combivent (4 mL) or saline solution (0.9% NaCl) (4 mL) will be administered once only to subjects.
  Other Names: Ipratropium - Salbutamol

SUMMARY:
Hypothesis: The reduction of dynamic hyperinflation and its negative effects on the respiratory system following a bronchodilator could lead to an improvement of cardiac function in terms of increased cardiac output. This may enhance oxygen delivery to the exercising muscles in COPD patients. Bronchodilator administration may also have an indirect effect on V'O2 kinetics via its action on cardiovascular and pulmonary variables.

Objectives:

1. To evaluate the effects of a bronchodilators on V'E , V'CO2 , and V'O2 kinetics in COPD during constant work-rate cycle exercise, and to evaluate whether bronchodilators will accelerate, indirectly, phase 2 kinetics (usually slower in COPD patients than normal subjects) and shorten t for V'E, V'CO2 , and V'O2 and shorten half-times for HR and O2 pulse, thus showing an improvement of oxygen transport to the peripheral active muscles.
2. To determine the impact of a bronchodilator-induced reduction in dynamic hyperinflation, and its effects on cardiovascular and pulmonary function, on exercise limitation in COPD.

DETAILED DESCRIPTION:
The inability to engage in the usual activities of daily living is one of the most distressing experiences of people afflicted with Chronic Obstructive Pulmonary Disease (COPD). Exercise intolerance progresses relentlessly as the disease advances and can lead to virtual immobility and social isolation. Our understanding of the complex interface between physiological impairment and disability in COPD has increased considerably in recent years. It has become clear that in COPD, exercise intolerance ultimately reflects integrated abnormalities of the ventilatory, cardiovascular, peripheral muscle and neurosensory systems. Ventilatory constraint is the dominant contributor to exercise limitation in more advanced disease. Recently, important studies have been conducted on the role of peripheral muscle dysfunction in exercise limitation in COPD.

The present study will test the hypothesis that the administration of bronchodilators (i.e., inhaled β2-agonist and inhaled anticholinergics in combination) in normoxemic COPD patients during moderate-intensity constant-load exercise may result in an enhancement of oxidative metabolism, reflected by reductions of O2 def and phase 2 tV'O2.

Fifteen normoxemic patients with stable COPD (FEV1 less than 60 % predicted) and severe chronic breathlessness (Baseline Dyspnea Index less than 6) will complete the study.

Each patient will perform three visits. At the first visit, patients will be familiarized with the various questionnaires and scales for rating the intensity and quality of symptoms and they will carry out pulmonary function testing and a symptom-limited incremental cycle exercise test in order to determine the anaerobic threshold (AT), the peak work-rate and the peak oxygen uptake. Each patient will subsequently complete two visits in which they will receive either nebulized bronchodilator (BD) (Combivent®, ipratropium 0.5 mg + salbutamol 2.5 mg) or placebo (PL), in random order. At 90-100 minutes post-dose, patients will perform pulmonary function tests, then they will perform a constant-load exercise test at 80% of AT V'O2. During constant-load exercise tests (2nd and 3rd visit), small samples of blood from the earlobe of each subject will be collected in order to determine the level of lactate and breathing gases (oxygen and carbon dioxide) in the blood.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years
* stable COPD
* FEV1 < 60 % predicted
* severe chronic breathlessness (Baseline Dyspnea Index < 6)

Exclusion Criteria:

* SpO2 at rest < 90% or a a sustained decrease of > 4% in arterial O2 saturation during the ergometer test, as determined by pulse oximetry
* a body mass index (BMI) < 19 or > 30
* chronic oral steroid therapy
* other medical conditions which could cause or contribute to breathlessness, i.e., heart disease or other respiratory diseases
* other problem which could interfere with carrying out of exercise testing, i.e., neuromuscular diseases, orthopedic diseases, etc.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
effects of bronchodilators on V'E , V'CO2 , and V'O2 kinetics in COPD during constant work-rate cycle exercise. | 2 hours post-inhalation of study drug
evaluate whether bronchodilators will accelerate, indirectly, phase 2 kinetics in COPD | 2 hours post-inhalation of study drug
evaluate whether bronchodilators will shorten t for V'E, V'CO2 , and V'O2 | 2 hours post-inhalation of study drug
evaluate whether bronchodilators will shorten half-times for HR and O2 pulse | 2 hours post-inhalation of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, Principal Investigator — Queen's University
Locations (1):
- Respiratory Investigation Unit (Queen's University), Kingston, Ontario, Canada

REFERENCES:
- [Derived] Laveneziana P, Palange P, Ora J, Martolini D, O'Donnell DE. Bronchodilator effect on ventilatory, pulmonary gas exchange, and heart rate kinetics during high-intensity exercise in COPD. Eur J Appl Physiol. 2009 Dec;107(6):633-43. doi: 10.1007/s00421-009-1169-4. Epub 2009 Aug 27. PMID 19711095